CLINICAL TRIAL: NCT05392829
Title: Reorientation of Tripped Patients 4 and 5 in Emergency Department to the City Medicine
Brief Title: Reorientation of Tripped Patients 4 and 5 in Emergency Department
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: CHSD_0016_URGENCES; 2021-A01989-32 (Other: IDRCB)
Record Dates: First submitted 2022-05-20; First posted 2022-05-26 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The increase in emergency room visits is partly related to the growing increase in unscheduled care, paradoxically associated with a decrease in the outpatient supply in the city. The "avoidable" passing rate is estimated at 43% in the last major DREES survey on hospital emergencies. Emergency services have been facing this challenge for years, but there is an urgent need to rethink its organizational model with the liberal system to meet this growing demand. Reorientation from the reception of emergencies is one of the avenues envisaged to face this challenge. It offers a different course from that of emergencies, provided that there are care structures equipped and adapted to unscheduled care. The Hospital in Saint-Denis is particularly faced with these challenges given a particular social ecosystem.

Methodology :

This single-center prospective observational study includes all adult patients sorted 4 and 5 by the reception organizing nurse, present during the survey.

The reorientation is one of the solutions proposed in the context of reorganizing access to care throughout the territory, appearing as one of the major public health issues in the coming years, it is appropriate to ask the question on a local scale. particularly exposed to the problem of unscheduled care, if patients are eligible for reorientation The non-medical factors identified as limiting the reorientation are: the absence of social cover, the language barrier, the patients referred by the samu or the fire brigade or a doctor, the patients who came by ambulance (because considered in theory as in the impossibility to move or having already been the subject of a "regulation")

Each 4 or 5 redirected patient is included and completes a questionnaire allowing the collection of information relating to their care pathways.

Primary endpoint :

Determine the proportion of patients not eligible for reorientation on non-medical criteria via a questionnaire, and identify the distribution of factors complicating reorientation

Secondary endpoints :

Identify the needs of patients re-orientated towards city medicine via the analysis of their passage to the emergency room, the reasons for their recourse to the emergency room (reasons, means and modes of arrival) their knowledge of the health system, and their relationship to general medicine

ELIGIBILITY:
Inclusion Criteria:

* patients tripped 4 and 5 at the IOA
* patients aged 18 years or older
* patients presenting to the emergency room every day of the week during the day and in the evening

Exclusion Criteria:

* patients triaged 1, 2, 3 at the IOA
* consulting patients for reasons requiring psychiatric advice
* unaccompanied minor patients
* patients brought by the police
* refusal or impossibility to participate
* protected adult patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years of age sorted 4 and 5 at the IAO present during the survey, at the hours of working days and the permanence of ambulatory care
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
socio-demographic characteristics | Day 1
  medical history, social security coverage, french language
reason for consultation | Day 1
  emergency assessment

SECONDARY OUTCOMES:
care pathway | Day 1
  time spent in the emergency room, additional examinations, diagnosic, becoming

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie GIRARD, Principal Investigator — Centre Hospitalier de Saint-Denis
Locations (1):
- Hôpital DELAFONTAINE, Saint-Denis, Île-de-France Region, France

REFERENCES:
- [Background] Guttmann A, Schull MJ, Vermeulen MJ, Stukel TA. Association between waiting times and short term mortality and hospital admission after departure from emergency department: population based cohort study from Ontario, Canada. BMJ. 2011 Jun 1;342:d2983. doi: 10.1136/bmj.d2983. PMID 21632665
- [Background] Marchetti M, Lepape M, Lauque D. La réorientation à l'accueil des services d'urgences : évaluation des pratiques professionnelles françaises. Ann Fr Médecine Urgence. 2014;4:349-353. doi:10.1007/s13341-014-0411-9
- [Background] Gilbert A, Brasseur E, Ghuysen A, D'Orio V. [New method to regulate unscheduled urgent care : the ODISSEE interactive self-triage platform]. Rev Med Liege. 2020 Mar;75(3):159-163. French. PMID 32157840
- See also: healthcare facilities 2020 — https://drees.solidarites-sante.gouv.fr/sites/default/files/2021-01/es2020.pdf
- See also: triage in emergency structure — https://www.sfmu.org/upload/referentielsSFMU/rfe_triage2013.pdf
- See also: ensuring first access to care — https://solidarites-sante.gouv.fr/IMG/pdf/rapport_snp_vf.pdf
- See also: National Survey of Hospital Emergency Structures, June 2013 — https://drees.solidarites-sante.gouv.fr/sources-outils-et-enquetes/01-enquete-nationale-sur-les-structures-des-urgences-hospitalieres-juin
- See also: survey and results DREES 2013 — https://drees.solidarites-sante.gouv.fr/sites/default/files/2020-08/er889.pdf
- See also: Information report by Mr. Philippe Boënnec tabled by the Delegation of the National Assembly for the Planning and Sustainable Development of the Territory on the permanence of care — https://www.assemblee-nationale.fr/13/rap-info/i1205.asp
- See also: health professionals as of January 1, 2018 — https://www.insee.fr/fr/statistiques/2012677